CLINICAL TRIAL: NCT03809416
Title: Combined Fractional LASERs Resurfacing With Platelets Rich Plasma (PRP) for Treating Post Acne Atrophic Scarring
Brief Title: Combined LASERs and PRP for Postacne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DEKA S.r.l. (Industry)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AY001
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Atrophic Acne Scar
Keywords: Acne scars; fractional lasers; PRP
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): 32 biopsy specimens from acne scars will be excised without any treatment.
- Lasers plus Normal Saline Solution (Sham Comparator): 32 biopsy specimens will be excised immediately after being treated with lasers and subsequent injection of normal saline solution.
  Interventions: Device: Lasers; Combination Product: Lasers plus Normal Saline Solution
- Lasers plus Platelets Rich Plasma (PRP) (Active Comparator): 32 biopsy specimens will be excised immediately after being treated with lasers and subsequent injection of platelets Rich Plasma (PRP).
  Interventions: Device: Lasers; Other: Platelets Rich Plasma

INTERVENTIONS:
Device: Lasers — Fractional carbon dioxide laser will be applied only over spots of deep post-acne scars, while Erbium: Glass will be applied all over face except to the two predetermined spots, i.e. control and another spot where NSS will be injected.
  Other Names: Fractional CO2 and Erbium Glass Lasers
  Arms: Lasers plus Normal Saline Solution; Lasers plus Platelets Rich Plasma (PRP)
Other: Platelets Rich Plasma — Platelet Rich Plasma (PRP) will be prepared from autologous blood collection in a syringe prefilled with anticoagulant solution followed by centrifugation then adding calcium gluconate 10% for induction of platelet activation. Activated PRP will be injected for all carbon dioxide laser spots in each patient immediately after each laser session except for two predetermined spots, i.e. control and sham comparator, which will be injected by normal saline solution (NSS).
  Other Names: PRP
  Arms: Lasers plus Platelets Rich Plasma (PRP)
Combination Product: Lasers plus Normal Saline Solution — Normal Saline Solution will be injected only in one spot after combined lasers resufacing to act as sham comparator compared to the other spot of Lasers plus PRP injection
  Other Names: NSS
  Arms: Lasers plus Normal Saline Solution

SUMMARY:
This study evaluates a new combined technique using two different laser wavelengths and Platelets Rich Plasma (PRP) to treat post-atrophic acne scars. Within the available knowledge of laser-tissue interactions and effects of PRP on wound healing, we will explore the clinical effects of our new combination procedure on a histopathological and immunohistochemical basis for guiding future post acne scars clinical research.

DETAILED DESCRIPTION:
The carbon dioxide and erbium lasers have been the gold and silver standards for acne scars treatment. As with selective photothermolysis, a major advance in the field is the incorporation of grids of MicroThermal Zones (MTZ) that spares islands of skin with an attractive treatment efficacy to downtime healing (5-7 days) ratio. Application of these fractionated resurfacing to carbon dioxide and erbium lasers allows deeper penetration into the skin.

Fractional photothermolysis was first described by as a new method for delivery of laser energy with the potential of laser safety and efficacy. Through the delivery of microscopic, non-contagious zones of thermal damage using a 1550 nm, mid-infra-red laser source, it was observed that surrounding islands of dermal and epidermal cells facilitated post-treatment collagen remodeling and rapid healing. Despite the success of minimally ablative and fractional technologies, there remained a need for more aggressive tissue ablation for the purposes of tissue rejuvenation of severely photodamaged skin and deeper rhytides. This might be due to the variability of architecture, depth, and width; thus, each type of scar has an optimal method by which it can be improved.

The idea of combining both carbon dioxide and erbium lasers appeared even before the era of fractional lasers. McDaniel et al, combined both non-fractional lasers for resurfacing of perioral rhytides comparing it to using carbon dioxide lasers alone and concluded that carbon dioxide laser resurfacing followed by 3 passes of erbium laser reduces the duration of crusting, swelling and itching when compared to carbon dioxide laser resurfacing alone with no significant difference in the outcome.

Later in 2010, the combination of fractional lasers carbon dioxide and erbium-doped laser was tried out for treating mild acne scars by a group of researchers. They reported a longer post laser erythema and hyperpigmentation, without precise pathogenesis. However, they suggested that these unexpected outcomes may have resulted from bulk heat damage to the surrounding tissues by heat stacking and recommended further studies to determine the optimal treatment parameters and reduce unexpected adverse reactions.

Platelet-rich plasma (PRP) is a high concentration of platelets in a small volume of plasma. PRP contains various growth factors and cytokines released by platelets, and those substances play a critical role in all aspects of the wound healing process. Among the stored mitogenic factors essential for wound repair are platelet-derived growth factor (PDGF) with the -AB and -C isoforms predominating, transforming growth factor β (TGF-β), vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), platelet-derived epidermal growth factor (PDEGF) and insulin-like growth factor-1 (IGF-1). These are variously involved in stimulating chemotaxis, cell proliferation, and maturation. PDGF is a powerful chemoattractant and stimulator of cell proliferation. All of them are potent angiogenic factors and endothelial cell mitogens. The wound healing effect of PRP is relatively well known, and PRP has been used in bone surgery, tendon and ligament repair, and chronic leg ulcer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with atrophic post-acne scars.
2. Patients without surgical &/or LASER resurfacing treatment for acne scars within the last 6 months.

Exclusion Criteria:

1. Pregnancy
2. Present or past history of hypertrophic scars or keloids
3. Present or past history of photosensitivity dermatoses including Connective Tissue Diseases.
4. Present history of herpes infection
5. Present history of Anemia (HGB < 10 g/dl), Thrombocytopenia &/or Platelets dysfunction.
6. Patients receiving isotretinoin within the last 3 months, NSAIDs within 72 hours of the procedure, anticoagulants &/or systemic use of corticosteroids within 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Patients' response denoting early Clinical improvement | 4 weeks after the 1st session
  calculating the change in 17 questions' responses of a new Patient Oriented Tool questionnaire for assessing Atrophic Acne Scarring through two parts; a) assessment of Acne Scar Appearance and b) Acne Scar Quality of Life questionnaire. Patients will record their responses before the 1st session and on the date of 2nd session.
Final Clinical improvement assessed using (0-10) scoring scale by blind assessors | 12 weeks after the 4th session
  The change in scores comparing 2 sets of digital photographs for each patient evaluated by 3 blind assessors, before and after 12 weeks of the 4th session. This blind assessment score will be compared to patients' score in their previous questionnaire.

SECONDARY OUTCOMES:
Higher new collagen formation in scars treated using lasers plus PRP technique | Immediately after the 1st session
  Picrosirus Red stained specimens under circularly polarized microscopy will be segmented into two color threshold bands (Green/Yellow G/Y and Red/Orange R/O) in the color HSB space. This will be numerically evaluated using ImageJ computer program
Immunohistochemical evaluation of Collagen I, Collagen III, and MMP-2 | Immediately after the 1st session
  Using a 4 grade scale (0, +, ++, +++), the 288 slides (i.e. 3 slides prepared from 96 specimens obtained from 32 patients) will be arranged for comparison among control, sham comparator and, active comparator. Also, results will be correlated to previous numerical ImageJ computerized assessment and patients' clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Lluis Puig, MD, PhD, Study Director — Universitat Autonoma de Barcelona (UAB); Alberto Calligaro, MD, PhD, Principal Investigator — University of Pavia
Locations (2):
- DEKA M.E.L.A. S.r.l., Florence, Calenzano, Italy
- Cosmetic Surgery Clinic, Al Qādisīyah, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Layton A, Dreno B, Finlay AY, Thiboutot D, Kang S, Lozada VT, Bourdes V, Bettoli V, Petit L, Tan J. Erratum to: New Patient-Oriented Tools for Assessing Atrophic Acne Scarring. Dermatol Ther (Heidelb). 2016 Jun;6(2):235-6. doi: 10.1007/s13555-016-0107-8. No abstract available. PMID 27008237
- [Result] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Result] Cho SB, Lee SJ, Kang JM, Kim YK, Oh SH. Combined fractional laser treatment with 1550-nm erbium glass and 10 600-nm carbon dioxide lasers. J Dermatolog Treat. 2010 Jul;21(4):221-8. doi: 10.1080/09546630903089650. No abstract available. PMID 19603309
- [Result] Lee JW, Kim BJ, Kim MN, Mun SK. The efficacy of autologous platelet rich plasma combined with ablative carbon dioxide fractional resurfacing for acne scars: a simultaneous split-face trial. Dermatol Surg. 2011 Jul;37(7):931-8. doi: 10.1111/j.1524-4725.2011.01999.x. Epub 2011 Jun 2. PMID 21635618
- [Result] Prignano F, Campolmi P, Bonan P, Ricceri F, Cannarozzo G, Troiano M, Lotti T. Fractional CO2 laser: a novel therapeutic device upon photobiomodulation of tissue remodeling and cytokine pathway of tissue repair. Dermatol Ther. 2009 Nov;22 Suppl 1:S8-15. doi: 10.1111/j.1529-8019.2009.01265.x. PMID 19891690